CLINICAL TRIAL: NCT03140228
Title: Postoperative Sore Throat in Children: Comparison Between Two Supraglottic Devices, Ambu® AuraOnce™ Laryngeal Mask Airway (LMA) and I-Gel® in Children Undergoing Elective Lower Abdominal or Orthopedic Surgery.
Brief Title: Postoperative Sore Throat in Children: Comparison Between Two Supraglottic Devices, Ambu® AuraOnce™ Laryngeal Mask Airway (LMA) and I-Gel®.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dr. Malika Hameed, Resident Anaesthesiology, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4249-Ane-ERC-16
Record Dates: First submitted 2017-04-29; First posted 2017-05-04 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Laryngeal Masks; Pharyngitis; Minors; Anesthesia
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- I-Gel group (Experimental): I-gel will be used for maintenance of airway during general anaesthesia
  Interventions: Device: I-Gel
- LMA ambu auraonce group (Active Comparator): LMA ambu auraonce will be used for maintenance of airway during general anaesthesia
  Interventions: Device: LMA

INTERVENTIONS:
Device: I-Gel — I-gel is the single use supraglottic airway from intersurgical, UK (Intersurgical Ltd, Wokingham, Berkshire, UK) with an anatomically designed mask made of a gel like thermoplastic elastomer to fit over perilaryngeal and hypopharyngeal structures. It is designed to separate the gastrointestinal and respiratory tracts and also allow a gastric tube to be passed into the stomach.
  Arms: I-Gel group
Device: LMA — The AmbuAuraOnce (Ambu A/S, Ballerup, Denmark) is a supraglottic airway device with an inflatable cuff. It is a disposable device as well, but unlike I-gel, it does not feature a gastric channel.
  Arms: LMA ambu auraonce group

SUMMARY:
Sore throat is minor but well recognized complaint after receiving general anaesthesia. It is rated as 8th most undesirable outcome in postoperative period.It not only affects the patient's satisfaction but also can affect patient activities after leaving hospital.

Many factors can contribute to postoperative sore throat and the incidence has been found to vary with the method by which airway is managed.

The study is conducted to compare the severity and frequency of postoperative sore throat in children undergoing elective surgery following the use of AmbuAuraOnce LMA and I-Gel. The study will be done in children who are able to self-report the severity of sore throat.

This study will help us to determine which supraglottic device (I-gel vs. AmbuAuraOnce LMA) is better in terms of causing less complication spells of sore throat. The use of such device will not only reduce the severity and frequency of postoperative sore throat that may affect the activities of patient after leaving hospital but also will improve satisfaction level of patient and parents.

DETAILED DESCRIPTION:
OBJECTIVE:

The objective of our study is to assess the frequency and severity of postoperative sore throat by comparison between two supraglottic devices, AuraOnce Laryngeal Mask Airway (LMA) and I-gel in children undergoing elective lower abdominal or orthopedic surgery.

HYPOTHESIS: Use of I-gel in children undergoing elective lower abdominal or orthopedic surgery is associated with decrease frequency and severity of postoperative sore throat as compared to use of AuraOnce Laryngeal Mask Airway.

ELIGIBILITY:
Inclusion Criteria:

* 6 to 16 year old patients of both gender
* ASA (American Society of Anesthesiologists) I and ASA II patients
* Scheduled for elective lower abdominal surgery (inguinal hernia repair or circumcision) or orthopedic surgery (upper and lower limb) under General anesthesia.

Exclusion Criteria:

* Patients with risk of aspiration (incomplete NPO (Nil per oral), Gastroesophageal reflux disease, Congenital anatomic abnormalities of aero digestive tract, delayed gastric emptying, altered mental status)
* Difficult airway(difficult mask ventilation or difficult laryngoscopy, Cormack-Lehane grade more than 2 in patient history, trismus, limited mouth opening, trauma or mass)
* Children who are unable to self-report pain using a four-point categorical pain scale
* Refusal of the parent
* Refusal of the child to give assent
* Patients having pre-existing sore throat or symptoms of Upper respiratory tract infection.
* Obese children i.e. BMI for age percentile equal to or greater than the 95th percentile on BMI-for-age percentile growth charts.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of postoperative sore throat | 24 hours
  To assess the frequency and severity of postoperative sore throat by comparison between two supraglottic devices, AuraOnce Laryngeal Mask Airway (LMA) and I-gel in children undergoing elective lower abdominal or orthopedic surgery.
  * Postoperative Sore Throat: Constant pain or discomfort in the throat which is independent of swallowing postoperatively for 24 hours.
  * Severity of Sore throat: The severity of sore throat will be measured by a four-point categorical pain scale.
  Grading of severity is as follow:
  0 = no sore throat
  1. mild (complains of sore throat only on asking)
  2. moderate (complains of sore throat on his/her own)
  3. severe (change of voice or hoarseness, associated with throat pain).
  Chi-square test will be applied to compare frequency and severity of post-operative sore throat between two groups. P ≤ 0.05 will be considered as significant.

SECONDARY OUTCOMES:
Immediate complications | Immediately after removal of supraglottic device
  Frequency will be calculated for immediate complications which includes laryngospasm, stridor, coughing, aspiration etc.
Insertion time | 5 minutes
  time of insertion of supraglottic device
Ease of insertion | 5 minutes
  Ease of insertion
Total number of attempts | 5 minutes
  maximum three attempts
Oropharyngeal seal pressure | 5 minutes
  seal pressure

CONTACTS AND LOCATIONS:
Overall Officials: Malika H Dhanani, FCPS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

REFERENCES:
- [Background] Higgins PP, Chung F, Mezei G. Postoperative sore throat after ambulatory surgery. Br J Anaesth. 2002 Apr;88(4):582-4. doi: 10.1093/bja/88.4.582. PMID 12066737
- [Background] Mokhtar AM, Choy CY. Postoperative sore throat in children: comparison between proseal LMA and classic LMA. Middle East J Anaesthesiol. 2013 Feb;22(1):65-70. PMID 23833853
- [Background] Kim H, Lee JY, Lee SY, Park SY, Lee SC, Chung CJ. A comparison of i-gel and LMA Supreme in anesthetized and paralyzed children. Korean J Anesthesiol. 2014 Nov;67(5):317-22. doi: 10.4097/kjae.2014.67.5.317. Epub 2014 Nov 26. PMID 25473460
- [Background] Theiler LG, Kleine-Brueggeney M, Luepold B, Stucki F, Seiler S, Urwyler N, Greif R. Performance of the pediatric-sized i-gel compared with the Ambu AuraOnce laryngeal mask in anesthetized and ventilated children. Anesthesiology. 2011 Jul;115(1):102-10. doi: 10.1097/ALN.0b013e318219d619. PMID 21572318
- [Background] Beylacq L, Bordes M, Semjen F, Cros AM. The I-gel, a single-use supraglottic airway device with a non-inflatable cuff and an esophageal vent: an observational study in children. Acta Anaesthesiol Scand. 2009 Mar;53(3):376-9. doi: 10.1111/j.1399-6576.2008.01869.x. PMID 19243322
- [Background] Verghese C, Brimacombe JR. Survey of laryngeal mask airway usage in 11,910 patients: safety and efficacy for conventional and nonconventional usage. Anesth Analg. 1996 Jan;82(1):129-33. doi: 10.1097/00000539-199601000-00023. PMID 8712387
- [Background] McHardy FE, Chung F. Postoperative sore throat: cause, prevention and treatment. Anaesthesia. 1999 May;54(5):444-53. doi: 10.1046/j.1365-2044.1999.00780.x. PMID 10995141